CLINICAL TRIAL: NCT04680949
Title: suPAR-Guided Anakinra Treatment for Validation of the Risk and Early Management of Severe Respiratory Failure by COVID-19: The SAVE-MORE Double-blind, Randomized, Phase III Confirmatory Trial
Brief Title: suPAR-Guided Anakinra Treatment for Management of Severe Respiratory Failure by COVID-19
Acronym: SAVE-MORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAVE-MORE
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Covid19
Keywords: SARS-CoV 2; anakinra
MeSH Terms: conditions — COVID-19 | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: The SAVE-MORE is a pivotal, confirmatory, phase III randomized clinical trial (RCT) aiming to evaluate the efficacy and safety of early start of anakinra guided by suPAR in patients with LRTI by SARS-CoV-2 in improving the clinical state of COVID-19 over 28 days as measured by the ordinal scale of the 11-point WHO clinical progression scale (CPS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients receiving standard-of-care (SOC) and placebo. Placebo is injected subcutaneously once daily for 10 days
  Interventions: Drug: Placebo
- Anakinra (Experimental): Patients receiving SOC and anakinra. Anakinra is injected subcutaneously as 100 mg once daily for 10 days
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Standard-of-care and anakinra. Anakinra is injected subcutaneously as 100 mg once daily for 10 days
  Other Names: Kineret
  Arms: Anakinra
Drug: Placebo — Standard-of-care and placebo. Placebo is injected subcutaneously once daily for 10 days
  Arms: Placebo

SUMMARY:
The SAVE-MORE is a pivotal, confirmatory, phase III randomized clinical trial (RCT) aiming to evaluate the efficacy and safety of early start of anakinra guided by suPAR in patients with LRTI by SARS-CoV-2 in improving the clinical state of COVID-19 over 28 days as measured by the ordinal scale of the 11-point World Health Organization (WHO) clinical progression scale (CPS).

DETAILED DESCRIPTION:
Since March 2020 when the COVID-19 pandemic started in Europe, the Hellenic Institute for the Study of Sepsis has launched in Greece the SAVE clinical trial (suPAR-guided Anakinra treatment for Validation of the risk and Early management of severe respiratory failure by COVID-19) (EudraCT number 2020-001466-11; approval 38/20 of the National Ethics Committee of Greece, approval IS 028/20 of the National Organization for Medicine of Greece, ClinicalTrials.gov identifier, NCT04357366). The concept of the SAVE trial was that early recognition of the risk for the progression of patients with lower respiratory tract infection (LRTI) by the new coronavirus SARS-CoV-2 into severe respiratory failure (SRF) may guide anakinra therapy to prevent SRF. The tool that was used for the diagnosis of risk for SRF is the biomarker suPAR (soluble urokinase plasminogen activator receptor) at measurable concentrations in the blood ≥6 ng/ml. The trial was designed to be open-label non-randomized and the idea was το the start of treatment well before any sign of respiratory failure emerges. Patients hospitalized at tertiary hospitals during the same time period as the SAVE trial was ongoing and who were receiving the same standard-of-care (SOC) treatment were studied as comparators. An interim analysis was submitted to the National Organization for Medicines; number 108002/23.10/2020. In this interim analysis, 130 patients receiving anakinra treatment and SOC were analysed and they were compared to 130 patients receiving SOC. The 130 SOC parallel comparators were selected by propensity score matching to be fully matched to the anakinra-treated patients for age, comorbidities, severity scores on the day of hospital admission, i.e. APACHE II score, Pneumonia Severity Index (PSI), Sequential Organ Failure Assessment (SOFA) and WHO severity, and for the intake of azithromycin, hydroxychloroquine and dexamethasone. SRF was defined as any respiratory ratio (pO2/FiO2) less than 150 mmHg necessitating mechanical ventilation or non-invasive ventilation (NIV). The results of this analysis may be summarized as follows:

* The incidence of SRF was significantly decreased from 59.2% in the parallel standard-of-care (SOC) comparators (n= 130) to 22.3% among the 130 anakinra-treated patients; hazard ratio, 0.30; 95% confidence intervals 0.20-0.46; P: 4.6 x 10-8.
* 30-day mortality was decreased from 22.3% in the SOC comparators to 11.5% among anakinra-treated patients; hazard ratio 0.49; 95% confidence intervals 0.25-0.97%; P: 0.041.
* Duration of stay at the intensive care unit was shortened with anakinra treatment compared to the SOC comparators for the patients who eventually developed SRF
* The median cost of hospitalization was significantly reduced from €2.398,40 among SOC comparators to €1.291,40 among anakinra-treated patients
* No safety concerns were raised.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or above 18 years
2. Male or female gender
3. In case of women, unwillingness to remain pregnant during the study period.
4. Written informed consent provided by the patient. For subjects without decision-making capacity, informed consent must be obtained from a legally designated representative following the national legislation in the Member State where the trial is planned.
5. Confirmed infection by SARS-CoV-2 virus
6. Findings in chest-X-ray or in chest computed tomography compatible with lower respiratory tract infection
7. Need for hospitalization for COVID-19. The need for hospitalization is defined by the attending physician taking into consideration clinical presentation, requirement for supportive care, potential risk factors for severe disease, and conditions at home, including the presence of vulnerable persons in the household.
8. Plasma suPAR ≥6ng/ml

Exclusion Criteria:

* Age below 18 years
* Denial for written informed consent
* Any stage IV malignancy
* Any do not resuscitate decision
* Αny pO2/FiO2 (partial oxygen pressure to fraction of inspired oxygen) ratio less than 150 mmHg irrespective if the patient is under mechanical ventilation (MV) / non-invasive ventilation (NIV) / extracorporeal membrane oxygenation (ECMO) or not
* Patient under MV or NIV or ECMO
* Any primary immunodeficiency
* Less than 1,500 neutrophils/mm3
* Plasma suPAR less than 6 ng/ml
* Known hypersensitivity to anakinra
* Oral or IV intake of corticosteroids at a daily dose equal or greater than 0.4 mg/kg prednisone for a period greater than the last 15 days.
* Any anti-cytokine biological treatment the last one month
* Severe hepatic failure defined as Child-Pugh stage of 3
* End-stage renal failure necessitating hemofiltration or peritoneal hemodialysis
* Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study
* Participation in any other interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the distribution of frequencies of each score of a 5-scale patient state evaluated from the 11-point WHO Clinical Progression ordinal Scale (CPS) between the two arms of treatment | 28 days
  Comparison of the distribution of frequencies of each score of the 5-scale patient state evaluated from the 11-point WHO Clinical Progression ordinal Scale (CPS) between the two arms of treatment by Day 28. This will be expressed as the distribution of the frequencies of each score of the scale in each arm of treatment by Day 28. The scale ranges from 0 (best outcome-asymptomatic) to 11 (worst outcome-death).

SECONDARY OUTCOMES:
Absolute change of the measure of the 11-point of WHO Clinical Progression ordinal Scale (CPS) | 28 days
  Comparison of the absolute change of the measure of the 11-point of WHO Clinical Progression ordinal Scale (CPS) between the two arms of treatment. The scale ranges from 0 (best outcome-asymptomatic) to 11 (worst outcome-death).
Relative change of the measure of the 11-point of WHO Clinical Progression ordinal Scale (CPS) | 28 days
  Comparison of the relative change (%) of the measure of the 11-point of WHO Clinical Progression ordinal Scale (CPS) between the two arms of treatment. The scale ranges from 0 (best outcome-asymptomatic) to 11 (worst outcome-death).
Absolute change of the measure of the 11-point of WHO Clinical Progression ordinal Scale (CPS) | 14 days
  Comparison of the absolute change of the measure of the 11-point of WHO Clinical Progression nordinal Scale (CPS) between the two arms of treatment. The scale ranges from 0 (best outcome-asymptomatic) to 11 (worst outcome-death).
Relative change of the measure of the 11-point of WHO Clinical Progression ordinal Scale (CPS) | 14 days
  Comparison of the relative (%) change of the measure of the 11-point of WHO Clinical Progression ordinal Scale (CPS) between the two arms of treatment. The scale ranges from 0 (best outcome-asymptomatic) to 11 (worst outcome-death).
Absolute change of the SOFA score | 14 days
  Comparison of the absolute change of the SOFA score (in points) between the two arms of treatment
Relative change of the SOFA score | 14 days
  Comparison of the relative (%) change of the SOFA score (in points) between the two arms of treatment
Absolute change of the SOFA score | 7 days
  Comparison of the absolute change of the SOFA score between the two arms of treatment
Relative change of the SOFA score | 7 days
  Comparison of the relative (%) change of the SOFA score between the two arms of treatment
Time until hospital discharge | 90 days
  Comparison of the time until hospital discharge between the two arms of treatment
Time until discharge from the intensive care unit | 90 days
  Comparison of the time until discharge from the intensive care unit between the two arms of treatment
Comparison of the rate of serious and non-serious adverse events between the two arms of treatment | 90 days
  Comparison of the rate of serious and non-serious adverse events between the two arms of treatment
Comparison of the rate of serious and non-serious adverse events between the two arms of treatment | 60 days
  Comparison of the rate of serious and non-serious adverse events between the two arms of treatment
Relative changes of circulating concentrations of suPAR (μg/liter), D-dimers (μg/liter), ferritin (μg/liter), and Interleukin-6 (μg/liter) by Day 7 from baseline Day 1 | 7 days
  Comparison of the relative changes of circulating concentrations of suPAR (μg/liter),D-dimers (μg/liter), ferritin (μg/liter), and Interleukin-6 (μg/liter) between the two arms of treatment
Relative changes of circulating concentrations of C-reactive protein (mg/liter) by Day 7 from baseline Day 1 | 7 days
  Comparison of the relative changes of circulating concentrations of C-reactive protein (mg/liter) between the two arms of treatment
Relative changes of circulating concentrations of suPAR (μg/liter),D-dimers (μg/liter), ferritin (μg/liter), and Interleukin-6 (μg/liter) by Day 4 from baseline Day 1 | 4 days
  Comparison of the relative changes of circulating concentrations of suPAR (μg/liter),D-dimers (μg/liter), ferritin (μg/liter), and Interleukin-6 (μg/liter) between the two arms of treatment
Relative changes of circulating concentrations of C-reactive protein (mg/liter) by Day 4 from baseline Day 1 | 4 days
  Comparison of the relative changes of circulating concentrations of C-reactive protein (mg/liter) between the two arms of treatment
Absolute change of the viral load by Day 7 from baseline Day 1 | 7 days
  Comparison of the absolute change of the viral load (in copies) between the two arms of treatment
Relative change of the viral load by Day 7 from baseline Day 1 | 7 days
  Comparison of the relative (%) change of the viral load between the two arms of treatment
Absolute change of the viral load by Day 4 from baseline Day 1 | 4 days
  Comparison of the absolute change of the viral load (in copies) between the two arms of treatment
relative change of the viral load by Day 4 from baseline Day 1 | 4 days
  Comparison of the relative change (%) of the viral load between the two arms of treatment
Transcriptomic analysis | 7 days
  Expression of messenger Ribonucleic Acid (mRNA) will be compared between the two arms of treatment
Proteomic analysis | 7 days
  Protein composition will be compared between the two arms of treatment

OTHER OUTCOMES:
Cost of hospitalization | 90 days
  Comparison of the cost of hospitalization between the two arms of treatment
Comparison of the distribution of frequencies of each score of a 5-scale patient state | 60 days
  Comparison of the distribution of frequencies of each score of the 5-scale patient state evaluated from the 11-point WHO Clinical Progression ordinal Scale (CPS) between the two arms of treatment by Day 28. This will be expressed as the distribution of the frequencies of each score of the scale in each arm of treatment by Day 60. The scale ranges from 0 (best outcome outpatients) to 5 (worst outcome-death)
Comparison of the distribution of frequencies of each score of a 5-scale patient state | 90 days
  Comparison of the distribution of frequencies of each score of the 5-scale patient state evaluated from the 11-point WHO Clinical Progression ordinal Scale (CPS) between the two arms of treatment by Day 28. This will be expressed as the distribution of the frequencies of each score of the scale in each arm of treatment by Day 90. The scale ranges from ) (best outcome-outpatients) to 5 (worst outcome-death)

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD, PhD, Study Chair — Hellenic Institute for the Study of Sepsis
Locations (40):
- Greece (32):
  - 2nd Department of Internal Medicine, University General Hospital of Alexandroupolis, Alexandroupoli
  - 10th Department of Pulmonary Medicine, SOTIRIA General Hospital of Chest Diseases of Athens, Athens
  - 1st Department of Internal Medicine, AMALIA FLEMING Prefecture General Hospital of Melissia, Athens
  - 1st Department of Internal Medicine, General Hospital of Athens KORGIALENIO-BENAKIO E.E.S., Athens
  - 1st Department of Internal Medicine, General Hospital of Eleusis THRIASIO, Athens
  - 1st Department of Internal Medicine, General Hospital of Nea Ionia CONSTANTOPOULIO-PATISION, Athens
  - 1st Department of Internal Medicine, General Hospital of Voula ASKLEPIEIO, Athens
  - 1st University Department of Internal Medicine, General Hospital of Athens LAIKO, Athens
  - 1st University Department of Pulmonary Medicine, SOTIRIA General Hospital of Chest Diseases of Athens, Athens
  - 2nd Department of Internal Medicine, General Hospital of Eleusis THRIASIO, Athens
  - 2nd Department of Pulmonary Medicine, SOTIRIA General Hospital of Chest Diseases of Athens, Athens
  - 2nd University Department of Internal Medicine, IPPOKRATEION General Hospital of Athens, Athens
  - 3rd Department of Internal Medicine, General Hospital of Athens KORGIALENEIO-BENAKEIO E.E.S., Athens
  - 3rd University Department of Internal Medicine, General Hospital of Chest Diseases of Athens SOTIRIA, Athens
  - 4th Department of Internal Medicine, ATTIKON University General Hospital, Athens
  - 4th Department of Pulmonary Medicine, SOTIRIA General Hospital of Chest Diseases of Athens, Athens
  - 5th Department of Pulmonary Medicine, SOTIRIA General Hospital of Chest Diseases of Athens, Athens
  - COVID-19 Department, General Hospital of Attica SISMANOGLEIO-AMALIA FLEMING, Athens
  - Department of Clinical Therapeutics, ALEXANDRA General Hospital of Athens, Athens
  - Department of COVID-19, Evangelismos General Hospital, Athens
  - Department of Internal Medicine, General Hospital of Athens Elpis, Athens
  - • 1st Department of Internal Medicine, General Hospital of Athens G. GENNIMATAS, Athens
  - • Department of Internal Medicine, General Hospital of Chest Diseases of Athens SOTIRIA, Athens
  - Department of Pulmonary Medicine, General Hospital of Kerkyra, Corfu
  - 1st Department of Internal Medicine, General University Hospital of Ioannina, Ioannina
  - Department of Internal Medicine, University General Hospital of Larissa,, Larissa
  - Department of Internal Medicine, University General Hospital of Patras PANAGIA I VOITHIA, Pátrai
  - 2nd Department of Internal Medicine, General Hospital of Piraeus TZANEIO, Piraeus
  - 1st Department of Internal Medicine, AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - 1st Department of Internal Medicine, PAPAGEORGIOU General Hospital of Thessaloniki, Thessaloniki
  - 2nd Department of Propedeutic Medicine, Ippokrateion University General Hospital of Thessaloniki, Thessaloniki
  - 3rd University Department of Internal Medicine, PAPAGEORGIOU General Hospital of Thessaloniki, Thessaloniki
- Italy (8):
  - Dipartimento di Medicina Dipartimento di Malattie Infettive, ASST Spedali civili, Brescia
  - Unità Operativa Clinica Malattie Infettive, Ospedale Policlinico San Martino, Genova
  - Dipartimento di Medicina Interna, Istituto Clinico Humanitas, Milan
  - Medicina Interna, Reumatologia, Immunologia, IRCCS San Raffaele, Milan
  - Dipartimento di Malattie Infettive e Tropicali e Microbiologia, IRCCS Ospedale Sacro Cuore Don Calabria, Negrar
  - Dipartimento di Malattie Infettive ad alta Intensità di cura ed altamente contagiose, IRCCS Lazzaro Spallanzani, Roma
  - Dipartimento Scienze di laboratorio e infettivologiche, Policlinico Universitario Agostino Gemelli, Roma
  - Dipartimento di Malattie infettive e tropicali-Università dell'Insubria, ASST dei Sette Laghi, Varese

REFERENCES:
- [Derived] Kyriazopoulou E, Kotsaki A, Safarika A, Poulakou G, Milionis H, Metallidis S, Adamis G, Fragkou A, Rapti A, Del Vecchio P, Kalomenidis I, Kitzoglou D, Angheben A, Kainis I, Iliopoulou K, Serino FS, Bakakos P, Tzavara V, Ioannou S, Dagna L, Dimakou K, Tzatzagou G, Chini M, Bassetti M, Kotsis V, Tsoukalas G, Selmi C, Nikolakopoulou S, Samarkos M, Doumas M, Masgala A, Papanikolaou I, Argyraki A, Akinosoglou K, Symbardi S, Panagopoulos P, Dalekos GN, Liesenfeld O, Sweeney TE, Khatri P, Giamarellos-Bourboulis EJ. 29-mRNA host response signatures for classification of bacterial infection, viral infection and disease progression in COVID-19 pneumonia: a post hoc analysis of the SAVE-MORE randomized clinical trial. Intensive Care Med Exp. 2025 Jun 30;13(1):67. doi: 10.1186/s40635-025-00777-1. PMID 40583075
- [Derived] Kyriazopoulou E, Hasin-Brumshtein Y, Midic U, Poulakou G, Milionis H, Metallidis S, Astriti M, Fragkou A, Rapti A, Taddei E, Kalomenidis I, Chrysos G, Angheben A, Kainis I, Alexiou Z, Castelli F, Serino FS, Bakakos P, Nicastri E, Tzavara V, Ioannou S, Dagna L, Dimakou K, Tzatzagou G, Chini M, Bassetti M, Kotsis V, Tsoukalas DG, Selmi C, Konstantinou A, Samarkos M, Doumas M, Masgala A, Pagkratis K, Argyraki A, Akinosoglou K, Symbardi S, Netea MG, Panagopoulos P, Dalekos GN, Liesenfeld O, Sweeney TE, Khatri P, Giamarellos-Bourboulis EJ. Transitions of blood immune endotypes and improved outcome by anakinra in COVID-19 pneumonia: an analysis of the SAVE-MORE randomized controlled trial. Crit Care. 2024 Mar 12;28(1):73. doi: 10.1186/s13054-024-04852-z. PMID 38475786
- [Derived] Akinosoglou K, Kotsaki A, Gounaridi IM, Christaki E, Metallidis S, Adamis G, Fragkou A, Fantoni M, Rapti A, Kalomenidis I, Chrysos G, Boni G, Kainis I, Alexiou Z, Castelli F, Serino FS, Bakakos P, Nicastri E, Tzavara V, Safarika A, Ioannou S, Dagna L, Dimakou K, Tzatzagou G, Chini M, Bassetti M, Kotsis V, Angheben A, Tsoukalas G, Selmi C, Spiropoulou OM, Samarkos M, Doumas M, Damoraki G, Masgala A, Papanikolaou I, Argyraki A, Negri M, Leventogiannis K, Sympardi S, Gatselis NK, Petrakis V, Netea MG, Panagopoulos P, Sakka V, Milionis H, Dalekos GN, Giamarellos-Bourboulis EJ. Efficacy and safety of early soluble urokinase plasminogen receptor plasma-guided anakinra treatment of COVID-19 pneumonia: A subgroup analysis of the SAVE-MORE randomised trial. EClinicalMedicine. 2023 Feb;56:101785. doi: 10.1016/j.eclinm.2022.101785. Epub 2022 Dec 26. PMID 36590789
- [Derived] Samaras C, Kyriazopoulou E, Poulakou G, Reiner E, Kosmidou M, Karanika I, Petrakis V, Adamis G, Gatselis NK, Fragkou A, Rapti A, Taddei E, Kalomenidis I, Chrysos G, Bertoli G, Kainis I, Alexiou Z, Castelli F, Saverio Serino F, Bakakos P, Nicastri E, Tzavara V, Kostis E, Dagna L, Koukidou S, Tzatzagou G, Chini M, Bassetti M, Trakatelli C, Tsoukalas G, Selmi C, Samarkos M, Pyrpasopoulou A, Masgala A, Antonakis E, Argyraki A, Akinosoglou K, Sympardi S, Panagopoulos P, Milionis H, Metallidis S, Syrigos KN, Angel A, Dalekos GN, Netea MG, Giamarellos-Bourboulis EJ. Interferon gamma-induced protein 10 (IP-10) for the early prognosis of the risk for severe respiratory failure and death in COVID-19 pneumonia. Cytokine. 2023 Feb;162:156111. doi: 10.1016/j.cyto.2022.156111. Epub 2022 Dec 14. PMID 36529030